CLINICAL TRIAL: NCT00310648
Title: Part 1:Phase I Open-Label, Single-Center to Evaluate the Safety of a Commercially Available Adjuvanted Influenza Vaccine When Administered to Elderly Subjects Part 2: A Phase III, Randomized, Controlled, Observer-Blind, Single-Center Study to Evaluate the Immunogenicity and Safety of a Commercially Available Influenza Vaccine and a Conventional Commercially Available Influenza Vaccine When Administered to Elderly Subjects
Brief Title: Comparative Trial Evaluating Safety and Immunogenicity of an Adjuvanted and a Conventional Influenza Vaccine in Elderly Subjects (> 60 Years)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry); Chiron s.r.l. Beijing Representative Office (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M70P1; Part 1: 200511-I; Part 2: 200511-III
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2006-09-14 (Estimated); Status verified 2006-09

CONDITIONS: Influenza
Keywords: Influenza, elderly, vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

INTERVENTIONS:
Biological: Influenza vaccine

SUMMARY:
Clinical Trial in Two parts:

Part 1: Phase I, Open-Label, Single-Center Study to Evaluate the Safety of an adjuvanted Influenza Vaccine When Administered to Elderly Subjects.

Part 2: A Phase III, Randomized, Controlled, Observer-blind, Single-Center Study to Evaluate the Immunogenicity and Safety of an adjuvanted and a conventional Influenza Vaccine When Administered to Elderly Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 60 years of age or older, mentally competent, willing and able to give the written informed consent prior to study entry

Exclusion Criteria:

* Any serious disease such as: cancer, autoimmune disease, advanced arteriosclerotic disease or complicated diabetes mellitus, chronic obstructive pulmonary disease (COPD) that requires oxygen therapy, acute or progressive hepatic disease, acute or progressive renal disease, congestive heart failure.
* Hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the vaccine.
* History of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine.
* Known or suspected (or have a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age).

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2006-01

PRIMARY OUTCOMES:
Requirements For Drug Registration & Guide Principles For ClinicaL Trial Techniques of Vaccine e.g Seroprotection, GMR's and Seroconversion rate at day 21 following vaccination.

SECONDARY OUTCOMES:
Solicited Local and Systemic Reactions Within 6 Days Following Vaccination And Adverse Events Thought the Study.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Drug Information Services, Study Director — Novartis Vaccines & Diagnostics
Locations (1):
- Nanning, Guangxi, China

REFERENCES:
- [Derived] Li R, Fang H, Li Y, Liu Y, Pellegrini M, Podda A. Safety and immunogenicity of an MF59-adjuvanted subunit influenza vaccine in elderly Chinese subjects. Immun Ageing. 2008 Feb 20;5:2. doi: 10.1186/1742-4933-5-2. PMID 18289372